# **Study Protocol**

**Title:** Effects of Topical Bromfenac Solution on Macular Thickness in Cataract Patients Undergoing Phacoemulsification Surgery

Clinical Trial Registration Number: NCT06785090

Document Date: March 28, 2025.

#### 1. Background and Rationale

Cystoid macular edema (CME) is a common postoperative complication following cataract surgery. Bromfenac, a topical nonsteroidal anti-inflammatory drug (NSAID), is hypothesized to reduce macular thickness and prevent CME. This study investigates the efficacy and safety of bromfenac in patients undergoing phacoemulsification.

## 2. Study Objectives

- **Primary Objective:** To assess the effect of bromfenac 0.09% ophthalmic solution on macular thickness after phacoemulsification.
- Secondary Objective: To evaluate potential adverse effects, including corneal erosion.

## 3. Study Design

- Study Type: Randomized controlled trial
- Allocation: Randomized
- Intervention Model: Parallel assignment
- **Masking:** Single-blinded (Investigator)

## 4. Eligibility Criteria

#### **Inclusion Criteria:**

- 1. All patients 18 years of age and older.
- 2. Patients diagnosed with cataracts.

#### **Exclusion Criteria**

- 1- Patients less than 18 years of age.
- 2- Patients with glaucoma, ocular hypertension, pseudo-exfoliation syndrome, or any optic nerve disease.
- 3- Patients with ocular diseases that might influence macular thickness, such as age-related macular degeneration, epiretinal membrane, history of uveitis, intraoperative complications, and traumatic cases.
- 4- Patients have undergone previous ocular surgery in the same eye, such as vitrectomy, intravitreal injection, retinal laser therapy, or corneal surgery
- 5- Patients who developed severe adverse effects from other drugs or had complications intraoperatively or postoperatively unrelated to bromfenac.
- 6- Patients take antiglaucoma medications.

- 7- Patients lost to follow-up.
- 8- Patients with an allergy to one of the postoperative medications.

## 5. Intervention and Follow-up

- **Group one** consisted of forty-five patients who received 0.09% bromfenac ophthalmic solution twice daily in addition to Moxifloxacin 0.5% ophthalmic drops every 6hrs and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6hrs.
- **Group two-** consisted of forty-two patients who received only Moxifloxacin 0.5% every 6hrs and Dexamethasone phosphate 0.1% ophthalmic drops every 4-6hrs without the administration of bromfenac 0.09% ophthalmic drops.

#### 6. Outcome Measures

- **Primary Outcome:** Change in central macular thickness (CMT) measured by Optical Coherence Tomography (OCT)
- Secondary Outcomes: adverse effects

#### 7. Statistical Methods

- Sample size calculation based on a power of 80% and significance level of 0.05.
- Independent t-test for intergroup comparisons.
- Paired t-test for intragroup pre- and post-treatment comparisons.

### **Statistical Analysis Plan (SAP)**

#### 1. Introduction

This SAP outlines the statistical methodologies for analyzing data collected in the clinical trial titled "Effects of Topical Bromfenac Solution on Macular Thickness in Cataract Patients Undergoing Phacoemulsification Surgery."

## 2. Study Population

- Intent-to-Treat (ITT) Population: All randomized patients.
- **Per-Protocol (PP) Population:** Patients who adhered to treatment and completed follow-up assessments.

#### 3. Statistical Methods

- **Descriptive Analysis:** Means and standard deviations (SD) for continuous variables.
- Inferential Analysis:

- **Primary Outcome:** Two-sample t-test for between-group comparisons of CMT change.
- Secondary Outcomes:
  - Incidence of CME: Chi-square test.
  - Adverse effects: Fisher's exact test.

## 4. Handling of Missing Data

- Missing data <5%: Complete case analysis.
- Missing data >5%: Multiple imputation methods.

## 5. Software Used

All analyses will be performed using SPSS.